CLINICAL TRIAL: NCT01127958
Title: DARE-Trial: Drug Eluting bAlloon for In-stent REstenosis. Multi-center, Randomized Trial to Study the Effect of the SeQuent Please Drug-eluting Balloon Versus the Xience Prime Drug-eluting Stent for the Treatment of In-stent Restenosis.
Brief Title: DARE-trial: A Trial Studying the Effect of the SeQuent Please Drug-eluting Balloon Compared to the Xience Prime Drug-eluting Stent for the Treatment of Stenosis of an Earlier Implanted Stent.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: B. Braun Medical B.V. (Industry)
Responsible Party: Principal Investigator, J. Baan, J. Baan, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL3148701810
Record Dates: First submitted 2010-05-18; First posted 2010-05-21 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: In-stent Restenosis
Keywords: In-stent restenosis; Minimal lumen diameter; Drug eluting balloon; Drug eluting stent
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SeQuent Please (Active Comparator): PCI with drug-eluting balloon
  Interventions: Device: PCI with a drug-eluting balloon
- Xience Prime (Active Comparator): PCI with a drug-eluting stent
  Interventions: Device: PCI with a drug-eluting stent

INTERVENTIONS:
Device: PCI with a drug-eluting balloon — PCI with a drug-eluting balloon for in-stent restenosis
  Arms: SeQuent Please
Device: PCI with a drug-eluting stent — PCI with a drug-eluting stent for in-stent restenosis
  Arms: Xience Prime

SUMMARY:
The main objective of the study is to determine whether PCI for in-stent restenosis with a drug eluting balloon is angiographically non-inferior to PCI with a drug eluting stent at 6 month follow up.

DETAILED DESCRIPTION:
Background of the study:

Coronary in-stent restenosis is commonly treated by using a drug eluting stent (DES). There are, however, some concerns about the safety of drug eluting stents, in particular with respect to delayed healing, chronic inflammatory reaction, and late or very late stent thrombosis. It is unknown whether the current treatment with another layer of stents may add to the risk of stent thrombosis or reoccurrence of restenosis. Therefore, the relatively new drug-eluting balloons may provide an alternative for treatment of in-stent restenosis, avoiding a double stent layer. The expected advantages of such drug-eluting balloons over stents are the ease of access of the lesion, the absence of a multiple stent layer, and the shorter necessity of the use of dual antiplatelet therapy. Several studies have demonstrated safety and efficacy of the Sequent Please drug-eluting balloon (DEB). Whether the drug eluting balloon is as effective as a drug eluting stent in preventing re-restenosis is not known.

Study design:

The study is designed as an multi-center, randomized, prospective two-arm trial with either PCI with a drug eluting balloon or a drug eluting stent for in-stent restenosis. Blinded evaluation of endpoints by independent core laboratory.

Study population:

The study population consists of 270 patients ( ≥ 18 years of age) with indication for PCI for in-stent restenosis of whom 135 are randomised to a drug eluting balloon and 135 are randomised to a drug eluting stent. Individuals have signed an informed consent for study measurements.

Intervention:

PCI with a drug-eluting stent, or PCI with a drug-eluting balloon.

ELIGIBILITY:
Inclusion Criteria:

* Restenosis of the initially stented main vessel, including ostial, left main and bifurcation lesions as well as venous or arterial grafts
* Restenosis of any type of stent; all drug-eluting stents or bare metal stents
* Restenosis must be present > 50% in-stent and < 5 mm out of the stent
* A reference diameter of ≥ 2.0 to 4.0 millimeters by visual estimation
* Amendable to PCI treatment with either the SeQuent ® Please DEB or the Xience™ Prime DES
* Amendable to dual antiplatelet treatment for the duration of 1 year
* Patients must be ≥ 18 years of age
* Patients must be able to understand the aim of the study, including risks, benefits and treatment alternatives
* Patients must agree to undergo a follow-up angiogram at 6 months (± 1 month)
* Patients must agree to undergo a clinical follow-up at 30 days, 6 months, 1, 2, 3, 4, and 5 years

Exclusion Criteria:

* The impossibility to arrange a follow-up coronary angiography at 6 months (± 1 month) after baseline procedure is considered an exclusion criterion for this study
* Patients have to meet the inclusion criteria;
* Life expectancy less than one year
* Severe renal insufficiency (glomerular filtration rate <30mL/min), with exception of of patients with renal dialysis
* STEMI
* Restenosis in a biodegradable stent
* Restenosis in a non CE marked stent
* Requirement for PCI in the same vessel or expected in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-05; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is the minimal lumen diameter (MLD) assessed by quantitative coronary angiography (QCA) at 6 months after PCI | 6 month's after PCI
  The primary objective of this study is to determine whether PCI with the SeQuent ® Please DEB versus PCI with the Xience™ Prime DES for the treatment of patients with in-stent restenosis is non-inferior with respect to minimal lumen diameter (MLD) assessed by quantitative coronary angiography (QCA) at six months.

SECONDARY OUTCOMES:
In-stent and in-segment percent Diameter Stenosis | 6 months
In-stent and in-segment Angiographic binary restenosis | 6 months
Persisting dissection (i.e. dissection post-index-procedure that remained present at follow-up), thrombosis and aneurysm | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Baan, Dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (8):
- Netherlands (8):
  - Academisch Medisch Centrum, Amsterdam
  - OLVG, Amsterdam
  - VUmc, Amsterdam
  - Tergooi Ziekenhuizen, Blaricum
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer ziekenhuis, Dordrecht
  - UMC St Radboud, Nijmegen
  - Isala klinieken, Zwolle